CLINICAL TRIAL: NCT00554684
Title: Treatment Intensity and Factors Predicting Short and Long Term Outcomes in Elderly and Very Elderly Patients Admitted to Intensive Care Units
Brief Title: Treatment Intensity/Factors Predicting Short and Long Term Outcomes in Elderly Critically Ill Patients
Status: Completed | Type: Observational
Sponsor: St. Luke's-Roosevelt Hospital Center (Other)
Responsible Party: Principal Investigator, Hassan Khouli, MD Director, Critical Care, St Luke's Roosevelt Hospital, St. Luke's-Roosevelt Hospital Center
Other Study IDs: 06-171
Record Dates: First submitted 2007-11-05; First posted 2007-11-07 (Estimated); Last update posted 2012-08-23 (Estimated); Status verified 2012-08

CONDITIONS: Critically Ill Very Elderly Patients Admitted to ICU's
Keywords: Outcome; Elderly; ICU; Quality of Life

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
1. Patients greater than 90 years of age will have poorer outcomes in terms of mortality than younger patients controlling for disease and acuity
2. Patients greater than 90 years old will consume more resources than younger patients controlling for disease and acuity
3. Patients greater than 90 years old will show lower levels of function than younger patients controlling for disease and acuity
4. Patients greater than 90 years old will show lower levels of HRQOL at 90-120 days post ICU discharge than younger patients controlling for disease and acuity

DETAILED DESCRIPTION:
Elderly patients make up between 26% and 51% of patients who are admitted to ICUs. The proportion of individuals in North America aged > 65 is projected to increase to 20% of the population by 2026. As population demographics change, and as new technologies, pharmaceuticals, and interventions prolong lives, the proportion of elderly patients admitted to ICUs and surviving ICU stay will continue to increase. Studies that have examined only ICU or hospital survival as an outcome have had variable results. Few studies have demonstrated that elderly ICU patients experience higher mortality rates, while others have demonstrated that age alone, when adjusted for other factors, is not an important prognostic indicator among elderly patients admitted to the intensive care units (ICU). However, age is still used as an important criteria for admission to ICUs. Most studies reviewed have looked at patients sixty-five to ninety years old. To our knowledge only two studies to date have addressed this issue among patients older than 90 to an ICU, both were retrospective.

With increasing age there is a parallel increase in health care costs. The use of expensive technology and procedures in the very elderly is fast becoming a major concern. Data on resource allocation and treatment intensity in the (90+) subgroup is sparse.

Beyond mortality and cost, health-related quality of life (HRQOL) is a fundamentally important end point of medical care. Few studies have addressed outcomes in terms of HRQOL and functional status of elderly following discharge the from critical care unit. These studies were limited by small number of subjects enrolled, retrospective design, and lack of validated tool to assess HRQOL.

We plan to prospectively collect data to look at determinants of treatment intensity, outcome, and resource allocation in elderly patients ages 65 and above admitted to the ICU with care taken to including as many patients in the age interval above 90 years of age. We will also assess HRQOL and functional status in very elderly patients who survive admission and are discharged from the hospital.

ELIGIBILITY:
Inclusion Criteria:

* Patients 65 year an older Admitted to MICU, SICU, and CCU

Exclusion Criteria:

* Patients who refuse to complete HRQL questionaire while hospitalized
* Subjects refuse to participate

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Critically Ill Elderly Patients
Sampling Method: Probability Sample
Enrollment: 399 (Actual)
Dates: Start 2007-07; Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hassan Khouli, MD, Principal Investigator — St. Luke's-Roosevelt Hospital Center
Locations (1):
- St. Luke's Roosevelt Hospital, New York, New York, United States